CLINICAL TRIAL: NCT06856941
Title: Cerebello-spinal Direct Current Stimulation Associated with Treadmill Gait Training in Functional Mobility in Patients with Parkinsons Disease
Brief Title: CsDCS on Functional Mobility in Parkinsons Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Doctor professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 78055423.8.1001.5208
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: gait training; parkinson disease; functional mobility; csDCS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- csDCS (Active Comparator)
  Interventions: Device: cerebello-spinal direct current stimulation
- csDCS sham (Sham Comparator)
  Interventions: Device: sham cerebello-spinal direct current stimulation

INTERVENTIONS:
Device: cerebello-spinal direct current stimulation — Cerebello-spinal direct current stimulation is an electrical stimulus in the cerebellum as well as in the spinal cord that is used to improve functional mobility. To our knowledge, this is the first study to use this setup in individuals with Parkinsons disease.
  Arms: csDCS
Device: sham cerebello-spinal direct current stimulation — Sham cerebello-spinal direct current stimulation involves masking, where the total duration of stimulation is thirty seconds, which is sufficient to mimic the sensation of stimulation but without neuromodulatory effects
  Arms: csDCS sham

SUMMARY:
Parkinsons disease is a progressive neurological disorder marked by a decline in the efficacy of dopaminergic synapses in the nigrostriatal pathway, causing motor disturbances. Resting tremor, bradykinesia, and muscle rigidity are the most prominent motor features. These factors result in gait impairments, including slowness and freezing. The primary treatment for the disease is medication. However, while medication does reduce motor symptoms, prolonged usage may lead to an increase of dyskinesias and a worsening of a patients clinical condition. Thus, alternative therapies, such as cerebellospinal direct current stimulation (csDCS), have gained popularity. Studies suggest that csDCS may be an effective approach to mitigate gait disorders in this patient population. Kinesiotherapy is an established therapeutic method that has been demonstrated to promote functional mobility and improve gait. To date, the combination of kinesiotherapy and csDCS has not been tested, thus the purpose of this study is to evaluate the effectiveness of this combined therapy for enhancing functional mobility in Parkinsons disease patients. The goal of this study is to assess the efficacy of blending csDCS and kinesiotherapy for improving patients functional mobility in Parkinsons disease. Two groups of volunteers will be assigned: i) actual csDCS + kinesiotherapy, and ii) sham csDCS + kinesiotherapy. The full procedure involves 10 therapy sessions conducted across two weeks.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of PD provided by a neurologist
* regular dopaminergic drug treatment (at least three months of use)
* aged 40 years or over
* staging I to IV on the modified Hoehn and Yahr scale

Exclusion Criteria:

* other neurological disorders, postural hypotension, vestibular, musculoskeletal or visual disorders that compromise performance in the proposed tests
* other osteoarticular diseases in the lower limbs that interfere with performance and locomotion
* a Montreal Cognitive Assessment (MoCA) score of less than 21 points
* have undergone previous surgery for PD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go | From enrollment to the end of treatment at 4 weeks
  For the TUG, the time taken by the patient to perform a task involving standing up from a chair, walking, and sitting back down is measured. The test begins with the patient seated in a chair with their back against the backrest. Upon request, the patient stands up, walks three meters at their fastest yet safe pace, turns around, returns to the chair, and sits down. Shorter times in completing this task indicate better functional mobility. Three repetitions of the test were recorded, and for analysis purposes, the average of the repetitions was used.

SECONDARY OUTCOMES:
Five times sit to stand test | From enrollment to the end of treatment at 4 weeks
  For the TSL5, the time taken by the patient to perform the task of sitting and standing from a chair five times consecutively is measured. The test begins with the patient seated in a chair with their back against the backrest. Upon request, the patient stands up and sits down five times at their fastest pace, but safely. Shorter times on this test indicate better functional mobility. The average of three attempts was used as the final result.
Mini balance evaluation system test | From enrollment to the end of treatment at 4 weeks
  The abbreviated version of the Balance Evaluation System Test (miniBESTest) assesses static and dynamic balance through six different balance control mechanisms based on 14 specific activities of daily living. Each activity is rated from 0 (worst performance) to 2 (best performance) points. Thus, lower scores indicate poorer balance.
Unified Parkinson Disease Rating Scale-II and Scale-III | From enrollment to the end of treatment at 4 weeks
  The motor function of the patients was assessed using the Unified Parkinsons Disease Rating Scale (UPDRS). The UPDRS is the most widely used clinical assessment tool for characterizing the motor symptoms of Parkinsons disease and for monitoring the progression of these symptoms and the physical disability caused by the disease. The UPDRS consists of 50 items, each rated from 0 to 4, ranging from the best (0) to the worst motor performance (4), and it is widely accepted for determining the efficacy of interventions in clinical studies. In the present study, Section II was used, which refers to the severity of the disease concerning the performance of activities of daily living. This section includes 13 items, each scored from 0 to 4, from the best to the greatest impairment. Section III of the UPDRS was also used, which corresponds to the motor examination and measures: resting tremor, postural tremor, rigidity, speech, facial expression, chair rise, posture, gait, postural stability
Freezing of gait questionnaire | From enrollment to the end of treatment at 4 weeks
  The Freezing of Gait Questionnaire (FOG-Q) is a scale that assesses the individual's subjective perception of the severity and impact of freezing on their gait performance. The FOG-Q is classified on a 5-point scale (0 to 4), with a total score ranging from 0 to 24. A higher score indicates that the individual's gait performance is more affected by freezing.
Six minute walking test | From enrollment to the end of treatment at 4 weeks
  In the 6MWT, the patient walks at their fastest, yet safe, pace along a 30-meter straight path for six minutes. At the end of the test, the total distance covered is calculated. Greater distances indicate better functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, Study Director — Universidade Federal de Pernambuco; João Fabrício, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided